CLINICAL TRIAL: NCT05906251
Title: An Open-Label, Systemic Gene Transfer Study to Evaluate the Safety, Tolerability, and Efficacy of SRP 6004 Administered by Systemic Infusion in Ambulatory Subjects With Limb Girdle Muscular Dystrophy Type 2B/R2 (LGMD2B/R2, Dysferlin Related)
Brief Title: A Gene Transfer Study to Evaluate the Safety, Tolerability and Efficacy of SRP-6004 in Ambulatory Participants With Limb Girdle Muscular Dystrophy, Type 2B/R2 (LGMD2B/R2, Dysferlin [DYSF] Related)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is being terminated due to a business decision.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-6004-102
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Limb Girdle Muscular Dystrophy
Keywords: Ambulatory; Gene-Delivery; LGMD2B/R2; Dysferlin; LGMD
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Limb-girdle muscular dystrophy, type 2B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-6004 (Experimental): Participants will receive single IV infusion of SRP-6004 on Day 1.
  Interventions: Genetic: SRP-6004

INTERVENTIONS:
Genetic: SRP-6004 — Single IV infusion of SRP-6004
  Other Names: rAAVrh74.MHCK7.DYSF.DV

SUMMARY:
The primary purpose of this study is to evaluate the safety of SRP-6004 administered by intravenous (IV) infusion in ambulatory participants with LGMD2B/R2 (DYSF related).

ELIGIBILITY:
Inclusion Criteria:

* Possess 1 homozygous or 2 heterozygous pathogenic and/or likely pathogenic DYSF Deoxyribonucleic acid (DNA) gene mutations as documented prior to screening visits.
* Participants must be ambulatory per protocol specified criteria.
* Ability to cooperate with motor assessment testing.
* Has accessible and intact lower and upper extremity musculature for biopsy.
* Have adeno-associated virus rhesus serotype 74 (rAAVrh74) antibody titers < 1:400 (that is, not elevated) as determined by enzyme-linked immunosorbent assay (ELISA).

Exclusion Criteria:

* Exposure to gene therapy, investigational medication, or other protocol-specified treatment within the protocol specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests.
* Presence of any other clinically significant illness, medical condition, or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risk for gene transfer.

Note: Other inclusion or exclusion criteria could apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious Adverse Events (SAEs) | Baseline up to Month 60

SECONDARY OUTCOMES:
Change from Baseline in Percent of Normal DYSF Protein Expression as Measured by Western Blot | Baseline, Day 90 and Month 15
Change from Baseline in Percent of Normal DYSF Protein Expression as Measured by Immunofluorescence (IF) Fiber Intensity | Baseline, Day 90 and Month 15
Change from Baseline in Percent of Normal DYSF Protein Expression as Assessed by IF Percent DYSF Positive Fibers (PPF: DYSF) | Baseline, Day 90 and Month 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States